CLINICAL TRIAL: NCT03599479
Title: The Efficacy of Virtual Reality Experiences on Acute Pain and Distress Caused by Fluoroscopic Pain Intervention in Chronic Pain Patients - A Randomized Controlled Clinical Trial
Brief Title: Virtual Reality Experiences on Acute Pain and Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Associate professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1802-028-920
Record Dates: First submitted 2018-06-24; First posted 2018-07-26 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Virtual Reality; Acute Pain; Anxiety
Keywords: Virtual reality; Acute pain; Anxiety
MeSH Terms: conditions — Acute Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Experimental): * After experiencing the VR machine in the transfer bed for 5 minutes, the subject moves to the operating room.
  * After the subject moves to the surgical bed, he/she takes the appropriate position for the fluoroscopic pain intervention, and wears the virtual reality device (headset, headphone, smartphone).
  * After the subject starts the VR program, the practitioner starts the fluoroscopic pain intervention.
  * Lidocaine skin infiltration and description of the practitioner during the intervention are performed with the intervention when necessary.
  Interventions: Device: Virtual reality group
- Conventional group (No Intervention): The fluoroscopic pain intervention is performed using only local anesthetics and description of the practitioner during the intervention as in the conventional cases.

INTERVENTIONS:
Device: Virtual reality group — Virtual reality group The study intervention is to provide acute pain management for the subject undergoing fluoroscopic pain intervention by using the virtual reality program provided by the collaborator through virtual reality device (headset, headphone, and smartphone) that are commercialized on the market.
  Other Names: Experimental
  Arms: Virtual reality group

SUMMARY:
The aim of this study is to evaluate the efficacy of virtual reality experiences on acute pain and distress caused by fluoroscopic pain intervention in chronic pain patient.

DETAILED DESCRIPTION:
The investigators perform lots of interventions for patients. But unfortunately, patients cannot help being exposed to the acute pain and fear during the interventions. "Virtual Reality(VR)" is a state-of-art advanced technology, which is now being extended to various medical fields such as pain management, dental treatment, body rehabilitation and cancer pain. There is no study that have conjugated the virtual reality experience for patients' acute pain and anxiety which occurs during the pain interventions. So the investigators like to evaluate the effects of virtual reality experience on acute pain and anxiety precipitated by the pain interventions.

ELIGIBILITY:
Inclusion Criteria:

If all of the following conditions are met :

* Patient who has chronic pain lasting more than 3 months and whose pain doctor determined that he or she needs following fluoroscopic pain intervention : Lumbar sympathetic ganglion block (LSGB), Fluoroscopic-guided pulsed radiofrequency ablation (pRF), Fluoroscopic-guided radiofrequency thermocoagulation (hRF)
* Adults who are at least 20 years of age
* Patients whose American Society of Anesthesiologists(ASA) physical status is classified as 1 or 2.
* A person who voluntarily agrees to participate in this clinical trial and has agreed in informed consent.

Exclusion Criteria:

If the subject falls under any of the following conditions :

* Patients who cannot have virtual reality experience due to hearing or visual impairment
* If the patient has difficulty communicating due to lack of cognitive ability
* Patients that examiners deemed unsuitable for this trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
11-point scale pain score | 15min after the procedure
  11-point scale pain score was assessed by the patient during the fluoroscopic-guided intervention, 0-10. 0 means no pain, 10 means the most severe pain one can imagine

SECONDARY OUTCOMES:
Hamilton Anxiety rating score (HAM-A) | 15min after the procedure
  total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Net Promotor Score (NPS) by patient | 15min after the procedure
  On a scale of 0 to 10, score 10 means most likely to recommend VR to a friend or a colleague
Net Promotor Score (NPS) by physician | 15min after the procedure
  On a scale of 0 to 10, score 10 means most likely to recommend VR to a friend or a colleague
Total amount of local anesthetics used to skin infiltration | intraoperative
  Total amount of local anesthetics used to skin infiltration (ml)
Total procedural time | intraoperative
  Total procedural time (minute)
Vital sign of the patient: Percutaneous oxygen saturation(SPO2,%) | Intraoperative
  Percutaneous oxygen saturation(SPO2,%)
Vital sign of the patient: noninvasive blood pressure(NIBP, mm Hg) | Intraoperative
  noninvasive blood pressure(NIBP, mm Hg)
Vital sign of the patient: electrocardiogram(ECG) | Intraoperative
  Arrhythmia
Vital sign of the patient: Heart rate (beat per minute) | Intraoperative
  Heart rate (beat per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youn Moon, MD, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linton SJ. A review of psychological risk factors in back and neck pain. Spine (Phila Pa 1976). 2000 May 1;25(9):1148-56. doi: 10.1097/00007632-200005010-00017. PMID 10788861
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307
- [Result] Hoffman HG, Patterson DR, Seibel E, Soltani M, Jewett-Leahy L, Sharar SR. Virtual reality pain control during burn wound debridement in the hydrotank. Clin J Pain. 2008 May;24(4):299-304. doi: 10.1097/AJP.0b013e318164d2cc. PMID 18427228
- [Result] Nilsson S, Finnstrom B, Kokinsky E, Enskar K. The use of Virtual Reality for needle-related procedural pain and distress in children and adolescents in a paediatric oncology unit. Eur J Oncol Nurs. 2009 Apr;13(2):102-9. doi: 10.1016/j.ejon.2009.01.003. Epub 2009 Feb 20. PMID 19230769